CLINICAL TRIAL: NCT01425671
Title: Neural Oscillations as Genetic and Functional Biomarkers in Normal and Disease States
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, L. Elliot Hong, L. Elliot Hong, University of Maryland, Baltimore
Other Study IDs: HP-00043082; R01MH085646 (NIH)
Record Dates: First submitted 2011-08-28; First posted 2011-08-30 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Family; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Schizophrenic patients, family members: Schizophrenia Spectrum Disorder Patients
- Controls: Normal controls

SUMMARY:
The principle aim of the project is to analyze brain electrical activity and genetic information that will help identify the nature and cause of the disease schizophrenia. This effort should lay the groundwork for future treatment in schizophrenic patients.

DETAILED DESCRIPTION:
There are several studies and hypotheses to be tested. This project includes a cross-sectional study design measuring brain waves, clinical symptoms, cognitive and functional ability, and genetic information in schizophrenic patients and normal controls. Subjects are expected to do a brain wave recording (EEG/ERP), role-play test designed to measure functionality and cognitive ability, and clinical symptom assessments. Expected duration of subject participation will be approximately 8 hours (about 2 visits). Outcome measures includes biomarkers, clinical symptoms and function, and genetic information.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female between ages 14-62 (clinical assessment and blood draw only above 62)
* Ability to give written assent (subjects who are below the age of 18)
* Ability to give written informed consent (age 18 or above)
* Sufficient understanding of the study and risks (ESC score 10 or above)
* Subjects above age 62 will not participate in brain electrical activity measurements although they may still participate in clinical assessments and blood draw.

Exclusion Criteria:

* Inability to sign informed consent/assent
* Any major medical illness that may affect normal brain functioning. Examples of these conditions include, but not limited to, stroke, repeated seizure, history of significant head trauma, CNS infection or tumor, an other significant brain neurological conditions.
* Significant alcohol or drug use (substance dependence within 6 months or substance abuse within 1 month) other than nicotine or marijuana dependence.
* Woman who is pregnant (child bearing potential but not on contraceptive and missing menstrual period; or by self-report; or by positive pregnancy test).
* Can not refrain from using alcohol and/or marijuana 24 hours or more& cigarette smoking half and hour or more prior to experiments.

Ages: 14 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Schizophrenic patients, family members, controls
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-11-30 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2024-01 (Actual)

PRIMARY OUTCOMES:
We will measure oscillatory abnormalities in resting, sensory response to single sound (SS), response to steady state auditory evoked potential , to a continuous matching task , and response during encoding and retrieval during a sensory retention task. | 10-12 hours

SECONDARY OUTCOMES:
Symptom and Cognition rating | 2 hrs

CONTACTS AND LOCATIONS:
Overall Officials: L.Elliot Hong, M.D., Principal Investigator — Maryland Psychiatric Research Center, Department of Psychiatry, University of Maryland School of Medicine
Locations (1):
- Maryland Psychiatric Research Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No